CLINICAL TRIAL: NCT03522090
Title: Retrospective Comparative Study of Routine Lower Neck CT in the Staging and Diagnosis of Lung Cancer Across Two Cohorts
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University College Hospital Galway (Other)
Collaborators: University Hospital Plymouth NHS Trust (Other)
Responsible Party: Principal Investigator, Mohammed Ahmed, Fellow in interventional respiratory medicine, University College Hospital Galway
Other Study IDs: V1.0
Record Dates: First submitted 2018-04-30; First posted 2018-05-11 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-04

CONDITIONS: Lung Cancer; Supraclavicular Lymphadenopathy
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- No neck CT: Cohort of patients with suspected lung cancer where the lower neck is not routinely included in CT
  Interventions: Diagnostic Test: lower neck CT
- Neck CT: Cohort of patients with suspected lung cancer where the lower neck is routinely included in CT
  Interventions: Diagnostic Test: lower neck CT

INTERVENTIONS:
Diagnostic Test: lower neck CT — Computerised tomography of the lower neck done as part of initial CT thorax and lower abdomen

SUMMARY:
This is a study comparing routine inclusion of the lower neck in initial CT thorax in patients with suspected lung cancer to not including it. The study aims to assess whether such an intervention reduces the number of invasive investigations required to achieve a final diagnosis and clinical stage and whether it improves the detection of cervical lymph nodes involvement by lung cancer.

DETAILED DESCRIPTION:
Two practices currently exist regarding the role of lower neck CT in patients with suspected lung cancer but with little evidence for either. Routine lower neck CT is potentially associated with benefits of higher detection of neck lymphadenopathy leading to better staging, less invasive procedure with positive implications for patients experience and care. The potential harms are delay in diagnosis due to false positive findings and radiation exposure. There is limited evidence in this area so this study will potentially provide evidence to inform health policy decisions based on the risk benefit balance.

This is a retrospective comparative study to assess the real-life impact of routine lower neck CT on the diagnostic and staging work up of patients with suspected lung cancer across two cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age > 18 years
* Pathologically confirmed primary lung cancer
* Intrathoracic N2 and or N3 disease on CT defined as lymph node with short diameter > 10 mm

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients initially seen with suspected lung cancer
Sampling Method: Non-Probability Sample
Enrollment: 164 (Estimated)
Dates: Start 2018-07-01 (Estimated); Primary Completion 2018-12-30 (Estimated); Study Completion 2019-01-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of pathologically confirmed malignant supraclavicular lymph node | 60 days from initial CT
  evidence of malignancy consistent with lung cancer on fine needle aspiration or core biopsy

SECONDARY OUTCOMES:
Number of diagnostic procedures performed per patient | 60 days from initial CT Thorax
  number of invasive procedures used to obtain tissue to achieve diagnosis and/or stage
Proportion of patients who underwent more than one diagnostic procedures | 60 days from initial CT Thorax
Proportion of patients who underwent Endobronchial Ultrasound (EBUS) | 60 days from initial CT Thorax

IPD SHARING:
Plan to Share IPD: No